CLINICAL TRIAL: NCT05332925
Title: Using Ex Vivo Tumoroids To Predict Immunotherapy Response In NSCLC (TUMORIN)
Brief Title: Using Ex Vivo Tumoroids To Predict Immunotherapy Response In NSCLC
Acronym: TUMORIN
Status: Recruiting | Type: Observational
Sponsor: Jun Zhang, MD, PhD (Other)
Collaborators: Nilogen Oncosystems (Industry)
Responsible Party: Sponsor-Investigator, Jun Zhang, MD, PhD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: IIT-2021-Tumorin
Record Dates: First submitted 2022-04-10; First posted 2022-04-18 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer; NSCLC; NSCLC Stage IV
Keywords: Tumoroids; Organoids; Immunotherapy; Immune check point inhibitor; Anti-PD-1; Anti-CTLA-4; Ex vivo model; 3D culture
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3-4 cores fresh tissue using 20g or larger core biopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Standard of care immune checkpoint inhbitors — This is NOT an interventional study.

SUMMARY:
To test whether it is feasible to perform the 3D-EX functional predictive response bioassay in the context of patients with advanced/metastatic NSCLC receiving immune checkpoint inhibitors in the standard of care clinical setting.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC), which accounts for approximately 85% of all lung cancer cases, remains the leading cause of cancer death worldwide. Immunotherapy such as using immune checkpoint inhibitors (ICIs) to target the programmed death-1 and its ligand (PD-1/L1) has revolutionized our management of this deadly disease.

However, a large proportion of patients do not derive benefit due to primary, adaptive or acquired resistance. Hence, better identifying this patient population, understanding the resistance mechanism and exploring novel combinations with current SOC immunotherapy are urgently needed to continue to benefit our NSCLC patients.

The investigators hypothesize that patient-derived immune cell containing ex-vivo tumoroids could serve these purposes. In this study, the investigators plan to develop such a 3D ex-vivo system utilizing fresh biopsied tissue from NSCLC patients. The investigators plan to prospectively evaluate the value of these ex-vivo tumoroids in immunotherapy naive advanced/metastatic NSCLC patients who will be receiving anti-PD-1/L1 (with or without anti-CTLA-4) per standard-of-care.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Patients with advanced/metastatic NSCLC
* Must be immunotherapy naive
* Males and females age ≥ 18 years
* ECOG Performance Status 0 - 2
* Measurable disease by RECIST 1.1
* Must have a lesion (either primary or metastatic lesion) that can be safely biopsied to have sufficient tissue (at minimum, 3-4 cores using 20g or larger core biopsy) to generate tumoroids
* Must have at least one target lesion to evaluate treatment response
* Will be receiving anti-PD-1/L1 with or without anti-CTLA-4 per standard of care Adequate organ function defined per standard of care in this setting.
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence or to use the forms of contraception as required/recommended by each immune checkpoint inhibitor used in the setting of standard of care.

Exclusion Criteria:

* Incarcerated
* Not competent to make medical decision, noncommunicative or noncompliant per investigator's judgement.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced/metastatic NSCLC patients who are immunotherapy naïve and ready to receive immune checkpoint inhibitors as standard--of-care treatment.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of establishing 3D ex-vivo tumoroid model | 2 years
  Twenty-five patients will be enrolled. The bioassay will be considered to be feasible if the 3D Ex-Vivo assay results are obtained on at least 20 patients.

SECONDARY OUTCOMES:
Correlation of response in ex vivo tumoroids with clinical objective response | 2 years
  To test whether the 3D-EX functional response bioassay can predict tumor response (using RECIST v1.1) in patients with advanced/metastatic NSCLC, receiving treatment with immune checkpoint inhibitors, in a standard clinical setting.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD, PhD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - The University of Kansas Cancer Center (KUCC), Fairway, Kansas
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas